CLINICAL TRIAL: NCT00128466
Title: Safety and Efficacy of Gentamicin Versus Streptomycin for the Treatment of Naturally Occurring Human Plague and Evaluation of Rapid Diagnostic Test Kits for Yersinia Pestis
Brief Title: Treatment and Diagnosis of Plague
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); Ministry of Health, Madagascar (Other Government); Ministry of Health, Uganda (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-3700
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Plague
Keywords: bubonic plague; pneumonic plague; septicemic plague; Yersinia pestis; Pasteurella pestis
MeSH Terms: conditions — Plague | interventions — Gentamicins; Streptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gentamicin
Drug: streptomycin

SUMMARY:
This clinical trial will compare the effectiveness of streptomycin, which historically is the standard drug for treatment of plague, with gentamicin. The hypothesis is that gentamicin is not inferior to streptomycin but that it will have less severe side effects. The study is being done in Madagascar because that country reports the most plague cases in the world. Patients coming into a participating clinic with suspected plague (bubonic, pneumonic, or septicemic) will be randomized into one of two treatment arms after giving informed consent. Patients will be monitored for side effects and for improvement of symptoms.

In addition, rapid diagnostic test strips have been developed but not fully evaluated for use on humans. The investigators will evaluate these new tests on specimens from the same patients, comparing their performance with that of classical diagnostic methods such as culture and serology.

DETAILED DESCRIPTION:
This protocol will guide clinical trials of treatment of naturally occurring human plague cases in African countries with a high incidence of human plague. The safety and efficacy of gentamicin will be compared to the standard drug regimen that is already used in Madagascar (streptomycin/co-trimoxazole) for treatment of plague. Data from this trial will be valuable to optimize clinical management of plague in many countries, including Madagascar and the United States.

In collaboration with the governments and health officials of Madagascar, the investigators will implement a randomized, controlled, non-blinded drug trial to compare the effectiveness and side effect profile of gentamicin to the national standard plague treatment.

Cases of plague will be identified through clinic-based surveillance in areas with a high incidence and/or in areas that have experienced outbreaks in recent years. After giving informed consent, patients will be randomly assigned to one of two treatment arms, each arm receiving a different antimicrobial. One patient group will be treated with gentamicin; the other group ("control group") will receive streptomycin alone or with co-trimoxazole.

This protocol will follow the national guideline of the Madagascar Ministry of Health, which means that patients with bubonic plague in the streptomycin treatment arm will receive streptomycin followed by trimethoprim-sulfamethoxazole. The only adaptation is that enrolled patients with renal insufficiency will receive adjusted dosing of streptomycin, whereas the national standard treatment does not call for dose adjustment in renal failure.

The investigators will also evaluate several newly available, rapid "dipstick" tests for the diagnosis of plague using serum, bubo aspirate, sputum, and urine specimens that will have already been collected from the patients enrolled in the drug trial. These rapid tests have been developed by several American companies and the Institut Pasteur in Madagascar, and have not been fully evaluated for use with human specimens. These results will be compared to standard diagnostic techniques. Such rapid diagnostic tests will be useful for plague diagnosis in developing nations and during bioterrorism events.

ELIGIBILITY:
Inclusion Criteria:

* 2 years of age or older.
* Patients must have had potential exposure to rodents and/or their fleas or contact with a known plague case.
* Patients must have a fever of at least 38 °C that developed rapidly, and have one of the following:

  * One or more buboes (defined as tender lymph node swelling >=1 cm) that appeared after or at the same time as the fever; or
  * Clinical suspicion of pneumonic plague (prostration, cough, increased respiratory rate, hemoptysis and/or purulent sputum); or
  * Clinical suspicion of plague AND an epidemiological link with other cases.
* Only patients that are later confirmed by standard diagnostic tests will be included in the final analysis. Patients who do not have plague confirmed by standard tests will still be included in the safety analysis.

Exclusion Criteria:

* Has signs fitting plague meningitis (severely ill patient with signs of plague and one or more of the following: headache, fever, sensorial disturbances, neck and back stiffness, and/or positive Kernig and Brudzinski signs).
* Has hypotension unresponsive to fluid therapy (i.e. shock). In adults hypotension is defined as systolic blood pressure < 80 mmHg and heart rate > 110/min; in children it will need to be diagnosed by attending physician or medical officer.
* Has an "illness severity score" of 16 or higher (see Patient Record)
* Has a known allergy to gentamicin, streptomycin, or trimethoprim-sulfamethoxazole
* Is receiving dialysis for renal failure
* Has other severe underlying disease such as hepatic failure or other severe organ failure
* Has taken tetracyclines, quinolones, gentamicin, streptomycin, trimethoprim-sulfamethoxazole, or chloramphenicol in the last 24 hours. If the patient has taken medications that are not known, he/she will still be enrolled.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-08; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Survival or death at 2 weeks

SECONDARY OUTCOMES:
Time to defervescence during treatment
Number and severity of adverse effects at 2 weeks
Complications at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Griffith, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Martin Schriefer, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Ministry of Health, Antananarivo, Antananarivo, Madagascar